CLINICAL TRIAL: NCT06429332
Title: International Care Bundle Evaluation in Cerebral Hemorrhage Research - a Batched Parallel Cluster-randomized Trial With a Baseline Period
Brief Title: International Care Bundle Evaluation in Cerebral Hemorrhage Research
Acronym: I-CATCHER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: The George Institute for Global Health, Australia (Other); Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-02523-01
Record Dates: First submitted 2024-05-14; First posted 2024-05-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-05

CONDITIONS: Intracerebral Hemorrhage; Intracerebral Haemorrhage; Intraventricular Hemorrhage; Stroke; Cerebrovascular Disease
Keywords: intracerebral hemorrhage; oral anticoagulant; blood pressure lowering; early intensive blood pressure lowering; care bundle; implementation study; reversal treatment; outcome; UW-mRS; Modified Rankin Scale
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Cerebrovascular Disorders | interventions — Resuscitation Orders; Standard of Care

STUDY DESIGN:
Intervention Model Description: international multicentre, batched, cluster. Patients are not randomized, hospitals will be randomized.
  In each batch, hospitals are randomized into two groups according to the timing of the intervention (Care Bundle) over 3 phases (usual care, randomized evaluation, post-implementation follow-up):
  Phase 1 - baseline routine data collection, training and formative study (assess context and local resources, support adjustment of the protocol into local pathways) Phase 2 - start intervention implementation in the intervention group, data collection for comparison with usual care in the control group Phase 3 - all hospitals implement the intervention, data collection for quality improvement, assess sustainability and integration
Who Masked: Outcomes Assessor
Masking Description: Treatment allocation is on a site-level and not on an individual level. The allocation is not blinded. Follow-up clinical outcome assessors, who have no prior association with the study and are unaware of the patients' allocation to either the intervention or control arm, will contact the participant by telephone at 6 months. At the initiation of contact, study subjects will be urged not to disclose their treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): A range of implementation methods will be used to introduce an active Care Bundle with time- and target-based metrics that involve the rapid correction of abnormal physiological variables over days or hospital discharge (or death, if sooner) and referral pathways
  Interventions: Other: Reversal of Oral anticoagulation within 30 minutes; Other: Early intensive blood pressure lowering; Other: Treatment of pyrexia; Other: Hyperglycemia treatment; Other: Do-not-resuscitate (DNR) or withdrawal of care; Other: Referral to Intensive Care; Other: Referral to Neurosurgery; Diagnostic Test: Repeat brain imaging
- Usual care (Placebo Comparator): For patients in the usual-care group, decisions about the location of care delivery, investigations, monitoring, and all treatments are made by the treating clinical team. Data will be collected regarding the management of patients, including insertion of invasive monitoring devices, intravenous fluid resuscitation, BP lowering, vasoactive support, glycemic control, mechanical ventilation, neurosurgery, and other supportive therapy.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Reversal of Oral anticoagulation within 30 minutes — In situations of either an elevated INR with the use of warfarin - treatment with either 3- or 4-factor prothrombin complex concentrate (PCC) or fresh frozen plasma (FFP) within 30 minutes of ICH diagnosis on NCCT to reach and maintain an INR target <1.3; or where there has been recent use (<48 hours) of a direct oral anticoagulant (DOAC), use of an appropriate reversal agent within 30 minutes, where available, and according to local approvals.
  Other Names: OAC reversal
  Arms: Intervention group
Other: Early intensive blood pressure lowering — A systolic blood pressure (BP) target of 130-140 mmHg within 30 minutes of ICH diagnosis on NCCT is strived for, and to maintain this BP level for the first 7 days (for patients presenting with blood pressure <200 mmHg). If blood pressure ≥200 and <220, a target BP of 160 mmHg should be targeted at 30 minutes, and 130-140 mmHg should be achieved in 60 minutes. If BP ≥220, target BP of 160 mmHg and should be achieved in 60 minutes.
  Arms: Intervention group
Other: Treatment of pyrexia — To achieve a body temperature target <37.5 °C within the first 24h following ICH diagnosis on NCCT
  Arms: Intervention group
Other: Hyperglycemia treatment — To maintain a blood glucose level 7-10 mmol/L within the first 24h following ICH diagnosis on NCCT
  Arms: Intervention group
Other: Do-not-resuscitate (DNR) or withdrawal of care — Refrain from the use of DNR or withdrawal of care orders for 48 hours
  Arms: Intervention group
Other: Referral to Intensive Care — Immediate (<30 min) referral to intensive care if airway, breathing and/or circulation are compromized
  Arms: Intervention group
Other: Referral to Neurosurgery — Immediate (<30 min) referral to neurosurgery if any of the following criteria are fulfilled:
  * Large and/or rapidly evolving supratentorial ICH (>20 ml volume)
  * Any intraventricular extension
  * Posterior fossa bleed, irrespective of volume
  * Suspicion of a vascular malformation, independent of volume or location
  * Reduction in reaction to sensory stimulation or drowsiness
  Arms: Intervention group
Diagnostic Test: Repeat brain imaging — Repeat 6-12-hour brain imaging with the physicians choice of modality, preferably computed tomography (CT), if clinical deterioration or the patient received OAC reversal treatment
  Arms: Intervention group
Other: Standard care — For patients in the usual-care group, decisions about the location of care delivery, investigations, monitoring, and all treatments are made by the treating clinical team. Data will be collected regarding the management of patients, including insertion of invasive monitoring devices, intravenous fluid resuscitation, BP lowering, vasoactive support, glycemic control, mechanical ventilation, neurosurgery, and other supportive therapy.
  Arms: Usual care

SUMMARY:
Spontaneous intracerebral haemorrhage (ICH) accounts for approximately 10-15% of all strokes but stands for 50% of stroke-related morbidity and mortality. Approximately half of all patients with ICH have a decreased level of consciousness at hospital admission. Despite this, intensive care and neurosurgical interventions are uncommon. A study conducted in low- and middle-income countries has demonstrated a beneficial effect of a treatment package consisting of early intensive blood pressure lowering, as well as the treatment of pyrexia and elevated blood glucose levels. The I-CATCHER team is now planning to conduct a similar study in Sweden and Australia, as well as in other high-income countries. The study has a clear focus on implementation, aiming to improve treatment and prognosis for patients with ICH within a few years. The purpose of I-CATCHER is to investigate whether a structured treatment package (Care Bundle) improves 3-month prognosis in patients with spontaneous ICH compared to standard care.

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage (ICH) accounts for 10 to 15% of all strokes in high-income countries (HIC), and nearly twice this number in low-income to upper-middle-income countries (LMIC) (29.5%). It is the most devastating type of stroke given the high one-month case fatality of approximately 30-40%, and only 12-39% suffer persistent disability.

Despite several advances in the management of acute ischemic stroke supported by numerous randomized controlled trials (RCT), progress in establishing novel interventions to improve outcomes for ICH has been slow. Still today, the diagnosis of ICH evokes pessimism among treating physicians, and patients may be withheld guideline adherent treatment for this reason. This nihilistic approach is presumably due to an over-estimation of poor outcome, often influenced by the neurologically devastating features commonly present at ICH admission. Additionally, the scarcity of RCTs providing strong evidence for treatment recommendations may contribute to a more reluctant approach in the acute setting of ICH, particularly when presenting with debilitating symptoms.

The third INTEnsive care bundle with BP reduction in acute cerebral hemorrhage trial (INTERACT3) was recently published in 2023. This trial employed a stepped wedge cluster RCT design to evaluate the implementation of a Care Bundle protocol. This comprehensive protocol included early intensive BP lowering (EIBPL), management of pyrexia and hyperglycemia, and the early reversal of OAC treatment. The design of this trial drew inspiration from a post-hoc analysis of the INTERACT2 study that showed that the scoring of abnormal baseline variables, interventions included in the future INTERACT3 Care Bundle, independently predicted a poor functional outcome following ICH. The implementation of the time sensitive bundle of care in INTERACT3 resulted in an improved functional outcome at 6 months following ICH. However, as the trial included patients predominantly from LMIC, further studies are warranted to determine if these results are applicable to HIC with a more applicable Care Bundle for these populations. An earlier intervention study from the United Kingdom, published in 2019, studied a similar 'quality improvement' acute Care Bundle. This Care Bundle aimed to improve the speed of treatment delivery, access to acute care, and decrease case fatality following ICH. Despite certain limitations, including a non-randomized design, this study demonstrated significantly lower mortality rates in patients receiving the Care Bundle versus the pre-implementation standard of care.

I-CATCHER is an international, multicenter, batched, parallel, cluster, randomized clinical trial (RCT) to assess a multifaceted package of protocols in a broad range of patients with acute ICH. In each batch, hospitals will be randomized into two groups according to the timing of the intervention (Care Bundle) over 3 phases (phase 1: usual care, phase 2: randomized evaluation - to intervention or usual care, phase 3: post-implementation follow-up - all hospitals implement the intervention). This design will capture consecutive patients with ICH and allow continued intervention in perpetuity as more hospitals join. Compared to a conventional stepped-wedge cluster RCT, the intervention effect in this design is less likely to be confounded by background temporal trends as only baseline and parallel comparison data (first 2 periods in bold black frame) are used to determine the effectiveness of the Care Bundle. All hospitals will be exposed to the Care Bundle which allows assessment of sustainability and integration of the intervention into routine practice. Each batch period is 18 months (6 months per phase); whole study will be rolled out in 2.5 years.

This design involves implementation of an intervention package applied to all patients with ICH as part of routine care. Patients are only excluded if they refuse to have details of their management included and/or participate in follow-up procedures.

Study site inclusion criteria: Organized systems of acute stroke care; no established comprehensive protocols for the management of ICH; suitable location, infrastructure and willingness to participate in clinical research; suitable numbers of ICH patients (at least 30 per year).

Patient inclusion criteria: Adults (≥18 years) with spontaneous ICH confirmed by imaging and admitted hospital within 24 hours of the onset of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years)
* Non-contrast computerized tomography (NCCT) imaging-verified diagnosis of spontaneous intracerebral haemorrhage
* ≤24 hours from symptom onset or presumed symptom onset (last seen well)

Exclusion Criteria:

* Previous care limitation
* End-stage comorbidity with short life-expectancy (<6 m; e.g. terminal cancer)
* ICH caused by brain tumor or cerebral venous thrombosis
* Clinical signs of brain herniation at first presentation (unresponsive patient with bilaterally fixed, maximally dilated pupils)
* Pregnant women beyond 22 weeks gestation may only be included after thorough discussion with an obstetrician to determine risks vs benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of functional outcome based on the Utility Weighted modified Rankin Scale score | 180±30 days
  The modified Rankin Scale (mRS) is an efficient, reliable, and simple functional outcome measure widely used as a primary endpoint in clinical trials for acute stroke. However, being an ordered categorical scale, it may not reflect potentially unequal differences in perceived quality of life associated with certain 1-point shifts vs others. Utility-weighted mRS is a score that weighs the mRS against a health utility scale, which defined as the desirability of a specific health outcome, facilitates comparisons of health-related quality of life across an array of clinical settings. Utility weights, as referred to hereafter, reflect the spectrum between perfect health (a score of 1) and outcomes worse than death (where death is a score of 0 and negative values indicate an outcome worse than death). The primary outcome is UW-mRS at 3 months and will be analyzed by means of a linear regression, with mRS as a dependent variable with 7 levels (0 [no residual symptom] to 6 [death]).

SECONDARY OUTCOMES:
Ordinal shift analysis of mRS | 180 days±30 days
  The assessment of shifts in the distribution of mRS scores through the evaluation of scores in ordinal groups
Assessment of health-related quality of life (HRQoL) | 180 days±30 days
  This will be assessed using the EuroQoL Group 5-Dimension self-report questionnaire (EQ-5D). The VAS is a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Poor outcome defined as mRS 3-6 | 180 days±30 days
  Binary secondary outcomes will be analyzed by means of standard GEE or random-effects regression with a logistic link and/or time-to-event type endpoints using the Cox model with a sandwich formula or a frailty model.
Separate outcomes for death and disability | 180 days±30 days
  Binary secondary outcomes will be analyzed by means of standard GEE or random-effects regression with a logistic link and/or time-to-event type endpoints using the Cox model with a sandwich formula or a frailty model.

CONTACTS AND LOCATIONS:
Locations (52):
- The University of Oklahoma Health, Oklahoma City, Oklahoma, United States
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Monash Medical Centre, Clayton
  - The George Institute for Global Health, Sydney
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada
- Hong Kong University Hospital, Hong Kong, Hong Kong
- Landspitali University Hospital, Reykjavik, Iceland
- Italy (5):
  - Avezzano Ospedale SS. Filippo e Nicola, Avezzano
  - Citta di Castello Ospedale Città di Castello, Città di Castello
  - Gubbio Ospedale di Gubbio e Gualdo Tadino, Gubbio
  - Azienda Ospedaliera Santa Maria della Misericordia Perugia, Perugia
  - Roma Policlinico Gemelli, Roma
- Malaysia (2):
  - National University of Malaysia Hospital, Kuala Lumpur
  - Universiti Putra Malaysia Hospital, Serdang
- Sweden (38):
  - Höglandssjukhuset i Eksjö, Eksjö
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Östra Sjukhuset, Gothenburg
  - Hässleholms Sjukhus, Hässleholm
  - Helsingborgs Lasarett, Helsingborg
  - Karolinska Universitetssjukhuset Huddinge, Huddinge
  - Länssjukhuset Ryhov, Jönköping
  - Länssjukhuset Kalmar, Kalmar
  - Blekingesjukhuset Karlskrona, Karlskrona
  - Blekingesjukhuset, Karlskrona
  - Centralsjukhuset Karlstad, Karlstad
  - Västmanlands sjukhus Köping, Köping
  - Centralsjukhuset Kristianstad, Kristianstad
  - Kungälvs sjukhus, Kungälv
  - Univeristetssjukhuset Linköping, Linköping
  - Ljungby Lasarett, Ljungby
  - Skåne University Hospital Lund Neurosurgery dept, Lund
  - Skåne University Hospital Lund, Lund
  - Region Skåne, Skåne University Hospital in Malmö, Department of Neurology, Malmo
  - Mölndals Sjukhus, Mölndal
  - Oskarshamn Sjukhus, Oskarshamn
  - Universitetssjukhuset Örebro, Örebro
  - Östersunds Lasarett, Östersund
  - Skaraborgs Sjukhus Skövde, Skövde
  - Capio St Görans Sjukhus, Stockholm
  - Södersjukhuset, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Danderyds sjukhus, Stockholm
  - Länssjukhuset Sundsvall, Sundsvall
  - Norra Älvsborgs Länssjukhus, Trollhättan
  - Norrlands Universitetssjukhus, Umeå
  - Lasarettet i Enköping, Uppsala
  - Akademiska Sjukhuset Uppsal, Uppsala
  - Hallands sjukhus Varberg, Varberg
  - Centrallasarettet Växjö, Vaxjo
  - Värnamo sjukhus, Värnamo
  - Västerås, Västerås
  - Ystads lasarett, Ystad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Draeger J, Wiezorrek R, Hock B, Gerhard E, Klemm M. [Physical technical calibration of a new self-tonometer]. Ophthalmologe. 1993 Feb;90(1):51-3. German. PMID 8443449
- [Background] Qureshi AI, Tuhrim S, Broderick JP, Batjer HH, Hondo H, Hanley DF. Spontaneous intracerebral hemorrhage. N Engl J Med. 2001 May 10;344(19):1450-60. doi: 10.1056/NEJM200105103441907. No abstract available. PMID 11346811
- [Background] van Asch CJ, Luitse MJ, Rinkel GJ, van der Tweel I, Algra A, Klijn CJ. Incidence, case fatality, and functional outcome of intracerebral haemorrhage over time, according to age, sex, and ethnic origin: a systematic review and meta-analysis. Lancet Neurol. 2010 Feb;9(2):167-76. doi: 10.1016/S1474-4422(09)70340-0. Epub 2010 Jan 5. PMID 20056489
- [Background] Parry-Jones AR, Sammut-Powell C, Paroutoglou K, Birleson E, Rowland J, Lee S, Cecchini L, Massyn M, Emsley R, Bray B, Patel H. An Intracerebral Hemorrhage Care Bundle Is Associated with Lower Case Fatality. Ann Neurol. 2019 Oct;86(4):495-503. doi: 10.1002/ana.25546. Epub 2019 Aug 16. PMID 31291031
- [Background] Hemphill JC 3rd, Newman J, Zhao S, Johnston SC. Hospital usage of early do-not-resuscitate orders and outcome after intracerebral hemorrhage. Stroke. 2004 May;35(5):1130-4. doi: 10.1161/01.STR.0000125858.71051.ca. Epub 2004 Mar 25. PMID 15044768
- [Background] Becker KJ, Baxter AB, Cohen WA, Bybee HM, Tirschwell DL, Newell DW, Winn HR, Longstreth WT Jr. Withdrawal of support in intracerebral hemorrhage may lead to self-fulfilling prophecies. Neurology. 2001 Mar 27;56(6):766-72. doi: 10.1212/wnl.56.6.766. PMID 11274312
- [Background] Zahuranec DB, Brown DL, Lisabeth LD, Gonzales NR, Longwell PJ, Smith MA, Garcia NM, Morgenstern LB. Early care limitations independently predict mortality after intracerebral hemorrhage. Neurology. 2007 May 15;68(20):1651-7. doi: 10.1212/01.wnl.0000261906.93238.72. PMID 17502545
- [Background] Logan JS, Bharucha H, Sloan JM. Mesotheliomas all: long before their time. Ulster Med J. 1996 May;65(1):1-2. No abstract available. PMID 8686093
- [Derived] Apostolaki-Hansson T, Ouyang M, Dowlatshahi D, Caso V, Bufi A, Law ZK, Billot L, Norrving B, Anderson CS, Ullberg T. International Care Bundle Evaluation in Cerebral Hemorrhage Research (I-CATCHER): Study protocol for a multicenter, batched, parallel, cluster-randomized trial with a baseline period. Int J Stroke. 2025 Aug;20(7):891-897. doi: 10.1177/17474930251342888. Epub 2025 May 12. PMID 40356012